CLINICAL TRIAL: NCT04872075
Title: Study on Prevention of SARS-CoV-2 Transmission During a Large Indoor Gathering Event
Acronym: SPRING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: PRODISS (Unknown); WEEZEVENT (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP210504; 2021-A01264-37 (Other: ID-RCB)
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Covid19
Keywords: Sars-Cov-2; Covid-19; Screening; Concert; Closed area; Standing configuration
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): People at the concert
  Interventions: Other: Concert; Diagnostic Test: Rapid nasopharyngeal antigen test for Sars-Cov-2; Diagnostic Test: Saliva Sample
- Control (Active Comparator): People staying at home
  Interventions: Diagnostic Test: Rapid nasopharyngeal antigen test for Sars-Cov-2; Diagnostic Test: Saliva Sample

INTERVENTIONS:
Other: Concert — People attending a concert in a closed area, with a mask
  Arms: Experimental
Diagnostic Test: Rapid nasopharyngeal antigen test for Sars-Cov-2 — A nasopharyngeal swab at inclusion (up to 3 days before concert) to confirm eligibility
Diagnostic Test: Saliva Sample — Saliva samples sent by participant at Day0 and Day7

SUMMARY:
The objective is to demonstrate if there is no increase in the risk of Sars-Cov-2 salivary carriage 7 days after a concert in the group participating in the event compared to a non participating group who stayed at home.

The hypothesis is that a systematic screening of Sars-Cov-2 within the 3 days before the event allows to control the risk of transmission and prevent cluster of transmission during the concert.

DETAILED DESCRIPTION:
Before inclusion, the participants will be able to pre-register to the event via a website. They will get an appointment for an inclusion visit at the Accor Arena (Paris Bercy, France).

During 3 days (from D-3 to D-1), participants with a registration will come to the Accor Arena to have a rapid Sars-Cov-2 antigen test (results in 15 min).

If the test is positive, the participant will be contacted and managed by the medical team in charge of the national strategy for positives cases.

People with a negative test will be included and randomized :

* Two kits with tube for collecting saliva samples (for D0 and D7) will be given to each participant at this visit
* People randomized in the experimental group will receive their concert ticket at a later date.
* At Day 0, people randomized in the experimental group, will come to the Accor Arena with their ticket to participate in the concert. At the entrance, they should give their D0 saliva sampling kit. The people randomized in the control group will stay at home and will send their D0 saliva sample by post mail.
* At Day 7 (±1 day) all the participants must return their D7 saliva sampling kit via post mail

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 45 years old
* lack of symptoms or no contact with people with Covid-19 in the last two weeks
* negative antigenic test to Covid-19 in the 3 days before the experiment
* people who declared to have no risk factor to severe form of Covid-19
* people who declared not to live in the same place as someone with these risk factors
* people residing in Ile-de-France area

Exclusion Criteria:

* positive test to Sars-Cov-2 within 3 days before the concert
* people with clinical signs suggesting infectious respiratory disease
* people with severe Covid-19 risk factor
* people living with someone having severe covid-19 risk factor
* not affiliated to social security
* people who cannot remain standing for the time of the experimentation (about 5 hours)
* person under tutorship or curatorship
* pregnant women or not having effective contraception method
* breastfeeding women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6678 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-06-13 (Actual); Study Completion 2021-06-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with a positive salivary RT-PCR at day 7 after the date of the concert | 7 days after the concert (-1/+8 days)
  Prove the lack of increase of salivary carriage risk of SARS-CoV-2 on day 7 in participants present at the concert (experimental group) compared to non-participants at the event (control group)

SECONDARY OUTCOMES:
Number of participants in each group with a positive salivary RT-PCR the day of the concert | The day of the concert
  Evaluation of the salivary carriage on day 0 (the concert day) despite a negative test within 3 days before the event and the conversion rate of salivary carriage between D0 and D7
Molecular analysis of transmission clusters | 7 days after the concert (-1/+8 days)
  Comparison of the sequence of complete viral genome in participant with a positive test at day 7
Average percentage of participants wearing their mask adequately for the duration of event | The day of the concert
  Estimate the overall compliance of the mask wearing by the participants during the duration of the event (covering nose and mouth)
Percentage of adequate mask wearing among participants according to location and time | The day of the concert
  Identify the circumstances (place, time) of failure of accurate mask wearing by the participants
Percentage of participants who downloaded and / or used the TousAntiCovid application at the time of inclusion | The day of the concert
  Estimate the feasibility and acceptability of using the Tousanticovid application

CONTACTS AND LOCATIONS:
Overall Officials: Constance DELAUGERRE, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AccorHotels Arena, Paris, France

REFERENCES:
- [Result] Delaugerre C, Foissac F, Abdoul H, Masson G, Choupeaux L, Dufour E, Gastli N, Delarue SM, Nere ML, Minier M, Gabassi A, Salmona M, Seguineau M, Schmitt S, Tonglet S, Olivier A, Poyart C, Le Goff J, Lescure X, Kerneis S, Treluyer JM; SPRING study group. Prevention of SARS-CoV-2 transmission during a large, live, indoor gathering (SPRING): a non-inferiority, randomised, controlled trial. Lancet Infect Dis. 2022 Mar;22(3):341-348. doi: 10.1016/S1473-3099(21)00673-3. Epub 2021 Nov 26. PMID 34843662